CLINICAL TRIAL: NCT06053216
Title: GuiDIng Energy Provision Using indiREct CalorimeTry: a Pilot Feasibility Randomised Controlled Trial in Critically Ill Adults With Obesity
Brief Title: Indirect Calorimetry Guided Energy Provision in Critically Ill Patients With Obesity
Acronym: DIRECT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Australian and New Zealand Intensive Care Research Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ANZIC-RC/OT001
Record Dates: First submitted 2023-08-21; First posted 2023-09-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Critical Illness; Obesity
Keywords: Critical care nutrition; Indirect calorimetry
MeSH Terms: conditions — Critical Illness; Obesity | interventions — Calorimetry, Indirect

STUDY DESIGN:
Intervention Model Description: A multi-centre, prospective, two arm parallel feasibility pilot randomised controlled trial
Masking Description: Open-label trial. However, clinicians will be blinded to indirect calorimetry measurements in the control arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Individualised energy delivery (Experimental): Energy delivery will be guided by indirect calorimetry, with the aim to meet 80-100% of the most recent energy expenditure measurement from day 4 to 28 of hospital admission.
  Interventions: Other: Indirect calorimetry
- Standard care nutrition (Active Comparator): Energy delivery will be according to predictive equation estimates and usual site practice from day 4 to 28 of hospital admission.
  Interventions: Other: Indirect calorimetry (Standard care nutrition arm)

INTERVENTIONS:
Other: Indirect calorimetry — Weekly indirect calorimetry measurements using the Q-NRG+ device will be used to guide energy delivery up to day 28 of hospital admission.
  Arms: Individualised energy delivery
Other: Indirect calorimetry (Standard care nutrition arm) — Weekly indirect calorimetry measurements using the Q-NRG+ device will be conducted up to day 28 of hospital admission. In the standard care nutrition arm, clinicians will be blinded to indirect calorimetry measurements.
  Arms: Standard care nutrition

SUMMARY:
The DIRECT trial is a prospective, multi-centre, two arm parallel feasibility pilot randomised controlled trial. The primary aim is to determine the feasibility of using repeat indirect calorimetry measurements to direct energy delivery in critically ill patients with obesity.

The trial will recruit 60 mechanically ventilated patients from 4-6 ICUs in Australia and New Zealand.

DETAILED DESCRIPTION:
Indirect calorimetry is the current reference standard for measuring energy expenditure during critical illness, allowing for personalisation of energy delivery. Use of indirect calorimetry may be important in mitigating under- and overfeeding and associated adverse outcomes. This may be particularly important in patients with obesity, where energy expenditure is difficult to estimate, and limited data is available on the optimal nutritional management of this subgroup.

Although access to indirect calorimetry is gradually improving, it remains an underutilised tool and skills required to complete and interpret measurements are limited which may hinder use and integration into practice. There is a resulting knowledge gap on the impact of indirect calorimetry on outcomes in comparison to standard care predictive equations.

A definitive and pragmatic trial is needed to assess the impact of guiding energy delivery with indirect calorimetry on patient outcomes. Importantly, confirming the feasibility of using indirect calorimetry to guide energy delivery is needed to define optimal measurement protocols prior to completion of a larger trial.

The primary aim of the DIRECT trial is to determine the feasibility of using repeat indirect calorimetry measurements to direct energy delivery in critically ill patients with obesity. The secondary aim is to inform a larger trial by collecting process, nutrition, functional, clinical and safety outcomes.

The investigators will consider the main trial feasible to conduct if 2 of the following 3 feasibility criteria are achieved: (a) recruitment rate is ≥ 1 patient per calendar month; (b) between group separation of ≥20% in energy adequacy during ICU admission is achieved in relation to measured energy expenditure and; (c) the number of indirect calorimetry measurements completed/planned ≥60% during ICU admission.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥ 18 years) patients
* Body mass index ≥30 kg/m2
* Between day 3 and 6 of index ICU admission
* Receiving invasive mechanical ventilation
* Receiving enteral or parenteral nutrition

Exclusion Criteria:

* Receiving extracorporeal membrane oxygenation support
* Major burns (≥20% total body surface area)
* Unable to perform indirect calorimetry within 24 hours of randomisation
* Known pregnancy
* Death is imminent
* Treating clinician believes the study is not in the best interest of the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-10-02 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Feasibility: Recruitment rate | During ICU admission (up to day 28)
  Patients per site, per month
Feasibility: Treatment separation in energy adequacy | During ICU admission (up to day 28)
  Energy adequacy % will be calculated as daily energy delivery (kcal)/ measured energy expenditure (kcal) and expressed as a percentage.
Feasibility: Protocol adherence | During ICU admission (up to day 28)
  Number of indirect calorimetry measurements completed/planned.

SECONDARY OUTCOMES:
Treatment separation in energy adequacy | Post-ICU period (up to day 28)
  Energy adequacy % will be calculated as energy delivery (kcal)/ measured energy expenditure (kcal) and expressed as a percentage
Protocol adherence | Post-ICU period (up to day 28)
  Number of indirect calorimetry measurements completed/ planned
Reasons for indirect calorimetry measurement non-completion | Up to day 28
  Reported overall and separately for ventilated and canopy measurements
Clinician acceptability relating to use of indirect calorimetry in routine clinical care (questionnaire) | Up to day 28
  Reported separately for ventilated and canopy measurements. A combination of yes/no, multiple-choice and Likert scale (1 (minimum) - 5 (maximum)) questions are included.
Patient acceptability relating to use of indirect calorimetry in routine clinical care (questionnaire) | Up to day 28
  Reported for canopy measurements only. A combination of yes/no, multiple-choice and Likert scale (1 (minimum) - 5 (maximum)) questions are included.
Cumulative difference in energy delivery compared to measured energy expenditure | Day 28
  kcal; reported overall and separately for ventilated and canopy measurements
Cumulative difference in energy delivery compared to prescribed energy expenditure | Day 28
  kcal; reported overall and separately for ventilated and canopy measurements
Nutritional status | Baseline, ICU (up to day 28) and hospital discharge (up to day 28)
  Assessed using the Global Leadership Initiative on Malnutrition (GLIM) criteria where malnutrition diagnosis is based on meeting predefined phenotypic and etiologic criteria (PMID: 30181091). Severity of malnutrition (moderate or severe) is determined based on the phenotypic criterion related to severity of unintentional weight loss.
Handgrip strength | Hospital discharge (up to day 28)
  Measured using a hand dynamometer
Duration of mechanical ventilation | Day 28
  Duration of mechanical ventilation (days)
ICU length of stay | Day 28
  Duration of ICU stay (days)
Hospital length of stay | Day 28
  Duration of hospital stay (days)
Survival | ICU discharge (up to day 28), in-hospital (up to day 28) and 90 day
  ICU, in-hospital and 90 day mortality
European Quality Of Life 5 Dimensions 5 Level (EQ5D-5L) | Day 90
  Health related quality of life assessment using EQ5D-5L. Each dimension has 5 levels ranging from no problems (1) to extreme problems (5), there is no overall score. It also has a visual analogue scale (VAS) ranging 0-100 with 0 being worst imaginable health state and 100 being best imaginable health state
World Health Organization Disability Assessment Schedule 2.0 (WHODAS) | Day 90
  WHODAS is a 12 point disability assessment with a raw score range of 0-48. 0 is no disability and 48 being full disability

CONTACTS AND LOCATIONS:
Locations (5):
- Australia (4):
  - Blacktown Hospital, Blacktown, New South Wales
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Ballarat Base Hospital, Grampians Health, Ballarat Central, Victoria
  - The Alfred Hospital, Melbourne, Victoria
- Department of Critical Care Medicine, Auckland City Hospital, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: Yes
Data sharing requests will be considered following publication of the primary trial data on an individual basis by the trial management committee (the data custodians). Data sharing will only be considered for investigator-initiated, independent researchers who provide a written data evaluation proposal that is judged to be methodologically sound. A data sharing agreement will be required to detail conditions under which data is shared and used. Resulting publications should appropriately cite and acknowledge the original data custodians. Requests for data sharing are to be made to anzicrc@monash.edu and the corresponding author, Dr Oana Tatucu; oana.tatucu@monash.edu